CLINICAL TRIAL: NCT00006030
Title: Protocol of a Randomized Trial for the Management of Small Well-Differentiated and Special Type Carcinomas of the Breast
Brief Title: Comparison of Four Different Treatment Regimens in Treating Women With Stage I Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: British Association of Surgical Oncology: Breast Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: BASO-BREAST-BASO-II; CDR0000068043 (Registry Identifier: PDQ (Physician Data Query)); EU-20019; ISRCTN47734678 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 2000-07-05; First posted 2004-03-25 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2006-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: tamoxifen citrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen by the tumor cells. Combining radiation therapy and tamoxifen with surgery may kill more tumor cells. It is not yet known which treatment regimen is most effective for stage I breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of four different treatment regimens in treating women who have stage I breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effectiveness of wide local excision alone versus wide local excision followed by radiotherapy with or without tamoxifen versus wide local excision plus tamoxifen in women with stage I breast cancer. II. Assess local occurrence in the treated breast, regional recurrence, distant recurrence, death from breast cancer, and occurrence of cancer in the opposite breast in these patients when treated with one of these regimens.

OUTLINE: This is a randomized study. Patients are randomized to one of four treatment arms. All patients undergo wide local excision of the tumor and axillary node dissection. Arm I: Patients undergo surgery only. Arm II: Patients undergo surgery followed by 25-35 radiotherapy treatments. Arm III: Patients undergo surgery plus oral tamoxifen daily for 5 years. Arm IV: Patients undergo surgery followed by 25-35 radiotherapy treatments and oral tamoxifen daily for five years. Patients are followed every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 1200 patients (300 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unilateral stage I invasive breast cancer No more than 1 tumor and no greater than 2 cm Grade 1 tumor of any histological type OR No special type OR Mixed type allowed No lymph node involvement No in situ carcinoma only or ductal carcinoma in situ with microinvasion No vascular invasion No Paget's disease of the nipple Well differentiated special type of primary mammary carcinoma including: Tubular Tubular/cribriform Cribriform Papillary Mucoid No lobular, medullary, or other rarer types of mammary carcinomas including: Adenoid cystic Carcinoid Secretory Spindle cell Apocrine No distant metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Under 70 Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing No other systemic disease that may preclude study No other prior malignancy except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: No other concurrent adjuvant systemic therapy

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-01

CONTACTS AND LOCATIONS:
Overall Officials: R.W. Blamey, Study Chair — Nottingham City Hospital
Locations (1):
- Nottingham City Hospital NHS Trust, Nottingham, England, United Kingdom